CLINICAL TRIAL: NCT01508026
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled, 8-Week Study to Evaluate the Safety and Efficacy of Nebivolol and Valsartan Given as a Fixed Dose Combination in Patients With Stage 1 or 2 Essential Hypertension
Brief Title: Study of the Efficacy and Safety of the Combination of Two FDA Approved Oral Medications, Nebivolol and Valsartan for Treatment of Stage 1 or 2 Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAC-MD-01
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-03

CONDITIONS: Stage 1 Hypertension; Stage 2 Hypertension
Keywords: Stage 1; Stage 2; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Nebivolol and Valsartan Fixed Dose Combination 1 (Experimental): Fixed Dose Combination Nebivolol 5 mg and Valsartan 80 mg
  Interventions: Drug: Nebivolol and Valsartan 1
- Nebivolol and Valsartan Fixed Dose Combination 2 (Experimental): Fixed Dose Combination Nebivolol 5 mg and Valsartan 160 mg
  Interventions: Drug: Nebivolol and Valsartan 2
- Nebivolol and Valsartan Fixed Dose Combination 3 (Experimental): Fixed Dose Combination Nebivolol 10 mg and Valsartan 160 mg
  Interventions: Drug: Nebivolol and Valsartan 3
- Nebivolol Low Dose (Experimental): Nebivolol Monotherapy 5 mg
  Interventions: Drug: Nebivolol 1
- Nebivolol High Dose (Experimental): Nebivolol Monotherapy 20 mg
  Interventions: Drug: Nebivolol 2
- Valsartan Low Dose (Experimental): Valsartan Monotherapy 80 mg
  Interventions: Drug: Valsartan 1
- Valsartan High Dose (Experimental): Valsartan Monotherapy 160 mg
  Interventions: Drug: Valsartan 2
- Placebo (Placebo Comparator): Dose Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nebivolol and Valsartan 1 — Fixed Dose Combination Nebivolol 5 mg and Valsartan 80 mg, oral administration, then dose doubled at Week 11 to Fixed Dose Combination Nebivolol 10 mg and Valsartan 160 mg, oral administration
  Arms: Nebivolol and Valsartan Fixed Dose Combination 1
Drug: Nebivolol and Valsartan 2 — Fixed Dose Combination Nebivolol 5 mg and Valsartan 160 mg, oral administration then dose doubled at Week 11 to Fixed Dose Combination Nebivolol 10 mg and Valsartan 320 mg, oral administration
  Arms: Nebivolol and Valsartan Fixed Dose Combination 2
Drug: Nebivolol and Valsartan 3 — Fixed Dose Combination Nebivolol 10 mg and Valsartan 160 mg, oral administration then dose doubled at Week 11 to Fixed Dose Combination Nebivolol 20 mg and Valsartan 320 mg, oral administration
  Arms: Nebivolol and Valsartan Fixed Dose Combination 3
Drug: Nebivolol 1 — Nebivolol Monotherapy 5 mg, oral administration, then dose doubled to at Week 11 to Nebivolol Monotherapy 10 mg, oral administration
  Arms: Nebivolol Low Dose
Drug: Nebivolol 2 — Nebivolol Monotherapy 20 mg, oral administration, then dose doubled to at Week 11 to Nebivolol Monotherapy 40mg, oral administration
  Arms: Nebivolol High Dose
Drug: Valsartan 1 — Valsartan Monotherapy 80 mg, oral administration, then dose doubled to at Week 11 to Valsartan Monotherapy, 160 mg, oral administration
  Arms: Valsartan Low Dose
Drug: Valsartan 2 — Valsartan Monotherapy 160 mg, oral administration, then dose doubled to at Week 11 to Valsartan Monotherapy, 320 mg, oral administration
  Arms: Valsartan High Dose
Drug: Placebo — Dose matched placebo, oral administration
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of fixed-dose combination of nebivolol and valsartan compared to monotherapy and placebo in patients with stage 1 and stage 2 hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients of age 18 years or above
* Patients diagnosed with stage 1 or stage 2 essential hypertension
* Normal physical examination findings, electrocardiogram (ECG) results and chest x-ray; or abnormal findings judged by the Investigator to be not clinically significant

Exclusion Criteria:

* Secondary hypertension or severe hypertension
* Clinically significant cardiovascular disease or heart failure
* Clinical significant respiratory disease that would prohibit the use of a beta blocker
* A medical contraindication to discontinuing a current antihypertensive therapy
* History of Type 1 diabetes mellitus
* History of Severe Mental Illness except mild depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4161 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in Sitting Diastolic Blood Pressure (DBP) | from basline to Week 8

SECONDARY OUTCOMES:
Change in Sitting Systolic Blood Pressure (SBP) | from baseline to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: David B Bharucha, MD, PhD, FACC, Study Director — Forest Laboratories
Locations (413):
- United States (413):
  - Forest Investigative Site 1750, Birmingham, Alabama
  - Forest Investigative Site 1038, Birmingham, Alabama
  - Forest Investigative Site 1308, Birmingham, Alabama
  - Forest Investigative Site 1192, Birmingham, Alabama
  - Forest Investigative Site 1005, Birmingham, Alabama
  - Forest Investigative Site 1047, Foley, Alabama
  - Forest Investigative Site 1717, Gulf Shores, Alabama
  - Forest Investigative Site 1056, Mobile, Alabama
  - Forest Investigative Site 1719, Muscle Shoals, Alabama
  - Forest Investigative Site 1145, Glendale, Arizona
  - Forest Investigative Site 1703, Goodyear, Arizona
  - Forest Investigative Site 1757, Mesa, Arizona
  - Forest Investigative Site 1170, Phoenix, Arizona
  - Forest Investigative Site 1238, Phoenix, Arizona
  - Forest Investigative Site 1204, Phoenix, Arizona
  - Forest Investigative Site 1755, Phoenix, Arizona
  - Forest Investigative Site 1259, Phoenix, Arizona
  - Forest Investigative Site 1001, Phoenix, Arizona
  - Forest Investigative Site 1078, Scottsdale, Arizona
  - Forest Investigative Site 1225, Tempe, Arizona
  - Forest Investigative Site 1712, Tempe, Arizona
  - Forest Investigative Site 1089, Tempe, Arizona
  - Forest Investigative Site 1065, Tucson, Arizona
  - Forest Investigative Site 1340, Tucson, Arizona
  - Forest Investigative Site 1331, Tucson, Arizona
  - Forest Investigative Site 1290, Little Rock, Arkansas
  - Forest Investigative Site 1138, Little Rock, Arkansas
  - Forest Investigative Site 1371, Pine Bluff, Arkansas
  - Forest Investigative Site 1220, Searcy, Arkansas
  - Forest Investigative Site 1063, Buena Park, California
  - Forest Investigative Site 1743, Burbank, California
  - Forest Investigative Site 1006, Carmichael, California
  - Forest Investigative Site 1384, Chino, California
  - Forest Investigative Site 1190, Chula Vista, California
  - Forest Investigative Site 1178, Costa Mesa, California
  - Forest Investigative Site 1043, Diamond Bar, California
  - Forest Investigative Site 1362, Encinitas, California
  - Forest Investigative Site 1144, Fresno, California
  - Forest Investigative Site 1095, Fresno, California
  - Forest Investigative Site 1710, Garden Grove, California
  - Forest Investigative Site 1022, Greenbrae, California
  - Forest Investigative Site 1370, Huntington Beach, California
  - Forest Investigative Site 1704, Huntington Park, California
  - Forest Investigative Site 1725, Huntington Park, California
  - Forest Investigative Site 1742, La Mesa, California
  - Forest Investigative Site 1381, Lomita, California
  - Forest Investigative Site 1706, Long Beach, California
  - Forest Investigative Site 1248, Los Angelas, California
  - Forest Investigative Site 1785, Los Angelas, California
  - Forest Investigative Site 1029, Los Angeles, California
  - Forest Investigative Site 1361, Los Angeles, California
  - Forest Investigative Site 1102, Los Angeles, California
  - Forest Investigative Site 1054, Mission Hills, California
  - Forest Investigative Site 1386, Moreno Valley, California
  - Forest Investigative Site 1756, Newport Beach, California
  - Forest Investigative Site 1181, Northridge, California
  - Forest Investigative Site 1212, Orange, California
  - Forest Investigative Site 1101, Palm Springs, California
  - Forest Investigative Site 1014, Paramount, California
  - Forest Investigative Site 1150, Pismo Beach, California
  - Forest Investigative Site 1009, Riverside, California
  - Forest Investigative Site 1241, Roseville, California
  - Forest Investigative Site 1046, Sacramento, California
  - Forest Investigative Site 1193, Sacramento, California
  - Forest Investigative Site 1296, Sacramento, California
  - Forest Investigative Site 1716, Sacramento, California
  - Forest Investigative Site 1096, San Bernardino, California
  - Forest Investigative Site 1189, San Diego, California
  - Forest Investigative Site 1279, San Diego, California
  - Forest Investigative Site 1354, San Diego, California
  - Forest Investigative Site 1724, San Diego, California
  - Forest Investigative Site 1106, San Diego, California
  - Forest Investigative Site 1027, San Francisco, California
  - Forest Investigative Site 1017, San Marino, California
  - Forest Investigative Site 1158, San Ramon, California
  - Forest Investigative Site 1318, Santa Ana, California
  - Forest Investigative Site 1239, Spring Valley, California
  - Forest Investigative Site 1792, Stockton, California
  - Forest Investigative Site 1301, Sylmar, California
  - Forest Investigative Site 1066, Temecula, California
  - Forest Investigative Site 1729, Tustin, California
  - Forest Investigative Site 1783, Westlake Village, California
  - Forest Investigative Site 1162, Colorado Springs, Colorado
  - Forest Investigative Site 1270, Denver, Colorado
  - Forest Investigative Site 1711, Denver, Colorado
  - Forest Investigative Site 1013, Northglenn, Colorado
  - Forest Investigative Site 1400, Thornton, Colorado
  - Forest Investigative Site 1324, Bridgeport, Connecticut
  - Forest Investigative Site 1045, Cromwell, Connecticut
  - Forest Investigative Site 1059, Stamford, Connecticut
  - Forest Investigative Site 1072, Waterbury, Connecticut
  - Forest Investigative Site 1159, Boca Raton, Florida
  - Forest Investigative Site 1007, Bradenton, Florida
  - Forest Investigative Site 1042, Brandon, Florida
  - Forest Investigative Site 1702, Brooksville, Florida
  - Forest Investigative Site 1764, Clearwater, Florida
  - Forest Investigative Site 1182, Coral Gables, Florida
  - Forest Investigative Site 1249, Coral Gables, Florida
  - Forest Investigative Site 1221, Cutler Bay, Florida
  - Forest Investigative Site 1793, Daytona Beach, Florida
  - Forest Investigative Site 1266, Deerfield Beach, Florida
  - Forest Investigative Site 1100, DeFuniak Springs, Florida
  - Forest Investigative Site 1734, DeLand, Florida
  - Forest Investigative Site 1775, Doral, Florida
  - Forest Investigative Site 1378, Doral, Florida
  - Forest Investigative Site 1237, Edgewater, Florida
  - Forest Investigative Site 1068, Fort Lauderdale, Florida
  - Forest Investigative Site 1026, Fort Lauderdale, Florida
  - Forest Investigative Site 1330, Fort Lauderdale, Florida
  - Forest Investigative Site 1794, Gainsville, Florida
  - Forest Investigative Site 1261, Hallandale, Florida
  - Forest Investigative Site 1240, Hialeah, Florida
  - Forest Investigative Site 1260, Hialeah, Florida
  - Forest Investigative Site 1155, Hollywood, Florida
  - Forest Investigative Site 1233, Jacksonville, Florida
  - Forest Investigative Site 1253, Jacksonville, Florida
  - Forest Investigative Site 1264, Jacksonville, Florida
  - Forest Investigative Site 1256, Jacksonville, Florida
  - Forest Investigative Site 1077, Jupiter, Florida
  - Forest Investigative Site 1041, Kissimmee, Florida
  - Forest Investigative Site 1399, Kissimmee, Florida
  - Forest Investigative Site 1784, Miami, Florida
  - Forest Investigative Site 1364, Miami, Florida
  - Forest Investigative Site 1206, Miami, Florida
  - Forest Investigative Site 1397, Miami, Florida
  - Forest Investigative Site 1180, Miami, Florida
  - Forest Investigative Site 1396, Miami, Florida
  - Forest Investigative Site 1154, Miami, Florida
  - Forest Investigative Site 1788, Miami, Florida
  - Forest Investigative Site 1223, Miami, Florida
  - Forest Investigative Site 1707, Miami, Florida
  - Forest Investigative Site 1282, Miami, Florida
  - Forest Investigative Site 1297, Miami Springs, Florida
  - Forest Investigative Site 1708, New Port Richey, Florida
  - Forest Investigative Site 1176, North Miami Beach, Florida
  - Forest Investigative Site 1284, Oldsmar, Florida
  - Forest Investigative Site 1232, Opa-locka, Florida
  - Forest Investigative Site 1802, Orlando, Florida
  - Forest Investigative Site 1049, Orlando, Florida
  - Forest Investigative Site 1235, Orlando, Florida
  - Forest Investigative Site 1741, Ormond Beach, Florida
  - Forest Investigative Site 1003, Oviedo, Florida
  - Forest Investigative Site 1369, Palm Harbor, Florida
  - Forest Investigative Site 1079, Pembroke Pines, Florida
  - Forest Investigative Site 1053, Pembroke Pines, Florida
  - Forest Investigative Site 1055, Pembroke Pines, Florida
  - Forest Investigative Site 1161, Pembroke Pines, Florida
  - Forest Investigative Site 1166, Pembroke Pines, Florida
  - Forest Investigative Site 1224, Pembroke Pines, Florida
  - Forest Investigative Site 1075, Pembroke Pines, Florida
  - Forest Investigative Site 1368, Pinellas Park, Florida
  - Forest Investigative Site 1023, Plant City, Florida
  - Forest Investigative Site 1737, Ponte Vedra, Florida
  - Forest Investigative Site 1749, Port Orange, Florida
  - Forest Investigative Site 1069, Saint Cloud, Florida
  - Forest Investigative Site 1315, Saint Cloud, Florida
  - Forest Investigative Site 1739, South Miami, Florida
  - Forest Investigative Site 1243, St. Petersburg, Florida
  - Forest Investigative Site 1723, St. Petersburg, Florida
  - Forest Investigative Site 1730, St. Petersburg, Florida
  - Forest Investigative Site 1076, Tamarack, Florida
  - Forest Investigative Site 1032, Tampa, Florida
  - Forest Investigative Site 1302, Tampa, Florida
  - Forest Investigative Site 1120, Winter Haven, Florida
  - Forest Investigative Site 1281, Atlanta, Georgia
  - Forest Investigative Site 1745, Atlanta, Georgia
  - Forest Investigative Site 1080, Blue Ridge, Georgia
  - Forest Investigative Site 1236, Lilburn, Georgia
  - Forest Investigative Site 1389, Marietta, Georgia
  - Forest Investigative Site 1002, Marietta, Georgia
  - Forest Investigative Site 1390, Oakwood, Georgia
  - Forest Investigative Site 1333, Sandy Springs, Georgia
  - Forest Investigative Site 1332, Savannah, Georgia
  - Forest Investigative Site 1252, Snellville, Georgia
  - Forest Investigative Site 1353, Snellville, Georgia
  - Forest Investigative Site 1740, Stockbridge, Georgia
  - Forest Investigative Site 1173, Woodstock, Georgia
  - Forest Investigative Site 1018, Honolulu, Hawaii
  - Forest Investigative Site 1398, Blackfoot, Idaho
  - Forest Investigative Site 1727, Boise, Idaho
  - Forest Investigative Site 1387, Hayden Lake, Idaho
  - Forest Investigative Site 1004, Meridian, Idaho
  - Forest Investigative Site 1039, Nampa, Idaho
  - Forest Investigative Site 1790, Addison, Illinois
  - Forest Investigative Site 1093, Arlington Heights, Illinois
  - Forest Investigative Site 1747, Chicago, Illinois
  - Forest Investigative Site 1071, Chicago, Illinois
  - Forest Investigative Site 1752, Chicago, Illinois
  - Forest Investigative Site 1403, Hazel Crest, Illinois
  - Forest Investigative Site 1126, Morton, Illinois
  - Forest Investigative Site 1283, O'Fallon, Illinois
  - Forest Investigative Site 1091, Evansville, Indiana
  - Forest Investigative Site 1103, Evansville, Indiana
  - Forest Investigative Site 1147, Muncie, Indiana
  - Forest Investigative Site 1107, Augusta, Kansas
  - Forest Investigative Site 1345, Hutchinson, Kansas
  - Forest Investigative Site 1805, Lenexa, Kansas
  - Forest Investigative Site 1255, Mission, Kansas
  - Forest Investigative Site 1092, Newton, Kansas
  - Forest Investigative Site 1801, Crestview Hills, Kentucky
  - Forest Investigative Site 1366, Lexington, Kentucky
  - Forest Investigative Site 1770, Louisville, Kentucky
  - Forest Investigative Site 1177, Madisonville, Kentucky
  - Forest Investigative Site 1251, Baton Rouge, Louisiana
  - Forest Investigative Site 1215, Covington, Louisiana
  - Forest Investigative Site 1274, Eunice, Louisiana
  - Forest Investigative Site 1323, Metairie, Louisiana
  - Forest Investigative Site 1795, Metairie, Louisiana
  - Forest Investigative Site 1285, New Orleans, Louisiana
  - Forest Investigative Site 1779, New Orleans, Louisiana
  - Forest Investigative Site 1769, Auburn, Maine
  - Forest Investigative Site 1125, Baltimore, Maryland
  - Forest Investigative Site 1263, Baltimore, Maryland
  - Forest Investigative Site 1128, Lutherville, Maryland
  - Forest Investigative Site 1726, Haverhill, Massachusetts
  - Forest Investigative Site 1061, Hyannis, Massachusetts
  - Forest Investigative Site 1728, North Dartmouth, Massachusetts
  - Forest Investigative Site 1356, Watertown, Massachusetts
  - Forest Investigative Site 1336, Chelsea, Michigan
  - Forest Investigative Site 1097, Flint, Michigan
  - Forest Investigative Site 1165, Kalamazoo, Michigan
  - Forest Investigative Site 1337, Stevensville, Michigan
  - Forest Investigative Site 1768, Traverse City, Michigan
  - Forest Investigative Site 1064, Troy, Michigan
  - Forest Investigative Site 1025, Belzoni, Mississippi
  - Forest Investigative Site 1057, Jackson, Mississippi
  - Forest Investigative Site 1034, Olive Branch, Mississippi
  - Forest Investigative Site 1271, Picayune, Mississippi
  - Forest Investigative Site 1782, Kansas City, Missouri
  - Forest Investigative Site 1250, St Louis, Missouri
  - Forest Investigative Site 1326, Missoula, Montana
  - Forest Investigative Site 1028, Bellevue, Nebraska
  - Forest Investigative Site 1388, Fremont, Nebraska
  - Forest Investigative Site 1313, Fremont, Nebraska
  - Forest Investigative Site 1035, Omaha, Nebraska
  - Forest Investigative Site 1016, Omaha, Nebraska
  - Forest Investigative Site 1254, Omaha, Nebraska
  - Forest Investigative Site 1148, Omaha, Nebraska
  - Forest Investigative Site 1044, Henderson, Nevada
  - Forest Investigative Site 1052, Henderson, Nevada
  - Forest Investigative Site 1011, Las Vegas, Nevada
  - Forest Investigative Site 1376, Las Vegas, Nevada
  - Forest Investigative Site 1019, Las Vegas, Nevada
  - Forest Investigative Site 1807, Las Vegas, Nevada
  - Forest Investigative Site 1048, Las Vegas, Nevada
  - Forest Investigative Site 1709, Edison, New Jersey
  - Forest Investigative Site 1132, Haddon Heights, New Jersey
  - Forest Investigative Site 1141, Linden, New Jersey
  - Forest Investigative Site 1227, Paramus, New Jersey
  - Forest Investigative Site 1169, Trenton, New Jersey
  - Forest Investigative Site 1338, Union, New Jersey
  - Forest Investigative Site 1761, Albuquerque, New Mexico
  - Forest Investigative Site 1796, Brooklyn, New York
  - Forest Investigative Site 1151, Buffalo, New York
  - Forest Investigative Site 1021, Glen Falls, New York
  - Forest Investigative Site 1115, Rochester, New York
  - Forest Investigative Site 1040, Asheboro, North Carolina
  - Forest Investigative Site 1073, Burlington, North Carolina
  - Forest Investigative Site 1142, Cary, North Carolina
  - Forest Investigative Site 1733, Charlotte, North Carolina
  - Forest Investigative Site 1067, Charlotte, North Carolina
  - Forest Investigative Site 1342, Dunn, North Carolina
  - Forest Investigative Site 1088, Greensboro, North Carolina
  - Forest Investigative Site 1385, Greensboro, North Carolina
  - Forest Investigative Site 1309, Greensboro, North Carolina
  - Forest Investigative Site 1306, Hickory, North Carolina
  - Forest Investigative Site 1098, Hickory, North Carolina
  - Forest Investigative Site 1110, Lenoir, North Carolina
  - Forest Investigative Site 1272, Mooresville, North Carolina
  - Forest Investigative Site 1024, Raleigh, North Carolina
  - Forest Investigative Site 1789, Raleigh, North Carolina
  - Forest Investigative Site 1715, Salisbury, North Carolina
  - Forest Investigative Site 1123, Shelby, North Carolina
  - Forest Investigative Site 1081, Wilmington, North Carolina
  - Forest Investigative Site 1705, Wilmington, North Carolina
  - Forest Investigative Site 1319, Winston-Salem, North Carolina
  - Forest Investigative Site 1405, Winston-Salem, North Carolina
  - Forest Investigative Site 1778, Winston-Salem, North Carolina
  - Forest Investigative Site 1203, Akron, Ohio
  - Forest Investigative Site 1210, Canal Fulton, Ohio
  - Forest Investigative Site 1012, Cincinnati, Ohio
  - Forest Investigative Site 1721, Cincinnati, Ohio
  - Forest Investigative Site 1280, Cincinnati, Ohio
  - Forest Investigative Site 1798, Cincinnati, Ohio
  - Forest Investigative Site 1732, Cincinnati, Ohio
  - Forest Investigative Site 1718, Cincinnati, Ohio
  - Forest Investigative Site 1062, Cincinnati, Ohio
  - Forest Investigative Site 1050, Cincinnati, Ohio
  - Forest Investigative Site 1084, Cleveland, Ohio
  - Forest Investigative Site 1765, Columbus, Ohio
  - Forest Investigative Site 1395, Columbus, Ohio
  - Forest Investigative Site 1209, Delaware, Ohio
  - Forest Investigative Site 1201, Lyndhurst, Ohio
  - Forest Investigative Site 1246, Maumee, Ohio
  - Forest Investigative Site 1135, Mount Gilead, Ohio
  - Forest Investigative Site 1322, Perrysburg, Ohio
  - Forest Investigative Site 1231, Willoughby, Ohio
  - Forest Investigative Site 1713, Zanesville, Ohio
  - Forest Investigative Site 1195, Norman, Oklahoma
  - Forest Investigative Site 1184, Oklahoma City, Oklahoma
  - Forest Investigative Site 1305, Oklahoma City, Oklahoma
  - Forest Investigative Site 1759, Oklahoma City, Oklahoma
  - Forest Investigative Site 1392, Yukon, Oklahoma
  - Forest Investigative Site 1116, Ashland, Oregon
  - Forest Investigative Site 1379, Eugene, Oregon
  - Forest Investigative Site 1780, Eugene, Oregon
  - Forest Investigative Site 1108, Hillsboro, Oregon
  - Forest Investigative Site 1294, Portland, Oregon
  - Forest Investigative Site 1109, Bensalem, Pennsylvania
  - Forest Investigative Site 1291, Bensalem, Pennsylvania
  - Forest Investigative Site 1090, Broomall, Pennsylvania
  - Forest Investigative Site 1218, Carnegie, Pennsylvania
  - Forest Investigative Site 1163, Downington, Pennsylvania
  - Forest Investigative Site 1118, Erie, Pennsylvania
  - Forest Investigative Site 1171, Erie, Pennsylvania
  - Forest Investigative Site 1383, Holland, Pennsylvania
  - Forest Investigative Site 1720, Jenkintown, Pennsylvania
  - Forest Investigative Site 1207, Lansdale, Pennsylvania
  - Forest Investigative Site 1314, Norristown, Pennsylvania
  - Forest Investigative Site 1198, Penndel, Pennsylvania
  - Forest Investigative Site 1293, Philadelphia, Pennsylvania
  - Forest Investigative Site 1137, Pittsburgh, Pennsylvania
  - Forest Investigative Site 1247, Red Lion, Pennsylvania
  - Forest Investigative Site 1791, Tipton, Pennsylvania
  - Forest Investigative Site 1196, Upper Saint Clair, Pennsylvania
  - Forest Investigative Site 1172, Warminster, Pennsylvania
  - Forest Investigative Site 1278, West Chester, Pennsylvania
  - Forest Investigative Site 1375, Warwick, Rhode Island
  - Forest Investigative Site 1760, Charleston, South Carolina
  - Forest Investigative Site 1363, Charleston, South Carolina
  - Forest Investigative Site 1122, Columbia, South Carolina
  - Forest Investigative Site 1133, Greenville, South Carolina
  - Forest Investigative Site 1809, Greenville, South Carolina
  - Forest Investigative Site 1327, Greer, South Carolina
  - Forest Investigative Site 1127, Mt. Pleasant, South Carolina
  - Forest Investigative Site 1310, Murrells Inlet, South Carolina
  - Forest Investigative Site 1152, Pelzer, South Carolina
  - Forest Investigative Site 1114, Simpsonville, South Carolina
  - Forest Investigative Site 1149, Spartanburg, South Carolina
  - Forest Investigative Site 1113, Summerville, South Carolina
  - Forest Investigative Site 1806, Union, South Carolina
  - Forest Investigative Site 1185, Dakota Dunes, South Dakota
  - Forest Investigative Site 1753, Rapid City, South Dakota
  - Forest Investigative Site 1402, Bristol, Tennessee
  - Forest Investigative Site 1037, Chattanooga, Tennessee
  - Forest Investigative Site 1031, Clarksville, Tennessee
  - Forest Investigative Site 1074, Collierville, Tennessee
  - Forest Investigative Site 1033, Fayetteville, Tennessee
  - Forest Investigative Site 1763, Kingsport, Tennessee
  - Forest Investigative Site 1744, Knoxville, Tennessee
  - Forest Investigative Site 1358, Memphis, Tennessee
  - Forest Investigative Site 1082, Memphis, Tennessee
  - Forest Investigative Site 1094, Arlington, Texas
  - Forest Investigative Site 1245, Austin, Texas
  - Forest Investigative Site 1311, Austin, Texas
  - Forest Investigative Site 1174, Beaumont, Texas
  - Forest Investigative Site 1762, Boerne, Texas
  - Forest Investigative Site 1244, Bryan, Texas
  - Forest Investigative Site 1776, Carrollton, Texas
  - Forest Investigative Site 1205, Corpus Christi, Texas
  - Forest Investigative Site 1268, Corsicana, Texas
  - Forest Investigative Site 1213, Dallas, Texas
  - Forest Investigative Site 1228, Houston, Texas
  - Forest Investigative Site 1372, Houston, Texas
  - Forest Investigative Site 1777, Houston, Texas
  - Forest Investigative Site 1157, Houston, Texas
  - Forest Investigative Site 1360, Houston, Texas
  - Forest Investigative Site 1230, Houston, Texas
  - Forest Investigative Site 1774, Houston, Texas
  - Forest Investigative Site 1262, Irving, Texas
  - Forest Investigative Site 1229, Longview, Texas
  - Forest Investigative Site 1199, New Braunfels, Texas
  - Forest Investigative Site 1214, Plano, Texas
  - Forest Investigative Site 1129, San Antonio, Texas
  - Forest Investigative Site 1766, San Antonio, Texas
  - Forest Investigative Site 1797, San Antonio, Texas
  - Forest Investigative Site 1295, San Antonio, Texas
  - Forest Investigative Site 1167, San Antonio, Texas
  - Forest Investigative Site 1186, San Antonio, Texas
  - Forest Investigative Site 1257, San Antonio, Texas
  - Forest Investigative Site 1317, San Antonio, Texas
  - Forest Investigative Site 1758, San Antonio, Texas
  - Forest Investigative Site 1334, Sugar Land, Texas
  - Forest Investigative Site 1269, Tomball, Texas
  - Forest Investigative Site 1349, Waco, Texas
  - Forest Investigative Site 1015, Clinton, Utah
  - Forest Investigative Site 1187, Draper, Utah
  - Forest Investigative Site 1226, Draper, Utah
  - Forest Investigative Site 1086, Magna, Utah
  - Forest Investigative Site 1216, Ogden, Utah
  - Forest Investigative Site 1219, Orem, Utah
  - Forest Investigative Site 1328, Riverton, Utah
  - Forest Investigative Site 1771, Salt Lake City, Utah
  - Forest Investigative Site 1175, Salt Lake City, Utah
  - Forest Investigative Site 1197, Salt Lake City, Utah
  - Forest Investigative Site 1194, Salt Lake City, Utah
  - Forest Investigative Site 1202, South Jordan, Utah
  - Forest Investigative Site 1773, St. George, Utah
  - Forest Investigative Site 1786, Arlington, Virginia
  - Forest Investigative Site 1130, Arlington, Virginia
  - Forest Investigative Site 1020, Burke, Virginia
  - Forest Investigative Site 1343, Danville, Virginia
  - Forest Investigative Site 1164, Manassas, Virginia
  - Forest Investigative Site 1767, Norfolk, Virginia
  - Forest Investigative Site 1292, Petersburg, Virginia
  - Forest Investigative Site 1131, Suffolk, Virginia
  - Forest Investigative Site 1099, Virginia Beach, Virginia
  - Forest Investigative Site 1119, Port Orchard, Washington
  - Forest Investigative Site 1394, Seattle, Washington
  - Forest Investigative Site 1085, Spokane, Washington
  - Forest Investigative Site 1335, Walla Walla, Washington
  - Forest Investigative Site 1377, Charleston, West Virginia
  - Forest Investigative Site 1367, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Giles TD, Weber MA, Basile J, Gradman AH, Bharucha DB, Chen W, Pattathil M; NAC-MD-01 Study Investigators. Efficacy and safety of nebivolol and valsartan as fixed-dose combination in hypertension: a randomised, multicentre study. Lancet. 2014 May 31;383(9932):1889-98. doi: 10.1016/S0140-6736(14)60614-0. PMID 24881993